CLINICAL TRIAL: NCT01514188
Title: A Multicenter, Randomized, Open-Label Phase 2b Study to Investigate the Preliminary Efficacy and Safety of INNO-206 (Doxorubicin-EMCH) Compared to Doxorubicin in Subjects With Metastatic, Locally Advanced, or Unresectable Soft Tissue Sarcoma
Brief Title: Preliminary Efficacy and Safety of INNO-206 Compared to Doxorubicin in Advanced Soft Tissue Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ImmunityBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INNO-206-P2-STS-01
Record Dates: First submitted 2012-01-12; First posted 2012-01-23 (Estimated); Results first posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2013-09

CONDITIONS: Metastatic Soft Tissue Sarcoma; Locally Advanced Soft Tissue Sarcoma; Unresectable Soft Tissue Sarcoma
Keywords: sarcoma; soft-tissue sarcoma; Metastatic,locally advanced, or unresectable soft tissue sarcoma
MeSH Terms: conditions — Sarcoma; Neoplasm Metastasis | interventions — DOXO-EMCH; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Doxorubicin (Active Comparator)
  Interventions: Drug: Doxorubicin
- INNO-206 (Experimental)
  Interventions: Drug: INNO-206

INTERVENTIONS:
Drug: INNO-206 — INNO-206 administered at 350 mg/m2 (260 mg/m2 doxorubicin equivalent) intravenously (IV) on Day 1 every 21 days for up to 6 consecutive cycles
  Other Names: DOXO-EMCH
  Arms: INNO-206
Drug: Doxorubicin — Doxorubicin administered at 75 mg/m2 for up to 6 consecutive cycles.
  Arms: Doxorubicin

SUMMARY:
This is a phase 2b, randomized, open-label, prospective, multicenter study comparing treatment with INNO 206 to doxorubicin in subjects with metastatic, locally advanced, or unresectable soft tissue sarcomas who have not been previously treated with any chemotherapy except potentially as adjuvant or neoadjuvant chemotherapy, and no evidence of tumor recurrence has occurred for at least 12 months.

DETAILED DESCRIPTION:
One hundred five subjects will be enrolled and randomized 2:1 to receive either INNO-206 or doxorubicin. INNO-206 at a dosage of 350 mg/m2 (doxorubicin equivalents of 260 mg/m2) will be administered as a 30 minute IVI on Day 1 of each cycle to approximately 70 subjects. Doxorubicin (75 mg/m2) will be administered to approximately 35 subjects on Day 1 of each cycle. An individual cycle of therapy will be defined as a 3-week (21-day) period. Cycles will be repeated every 3 weeks. Multiple cycles may be administered until the subject is withdrawn from therapy or until a maximum of 6 cycles are administered. Overall response rates as well as individual categories of response (CR, PR, SD, and PD) will be determined using RECIST 1.1.[28] Time-to-event endpoints, including PFS and OS will be assessed using the Kaplan Meier method.[30] Evaluation of 4- and 6-month progression-free survival will also be performed. Toxicity (adverse events) will be recorded using the NCI CTCAE, version 4.0 (published 28 May 2009).

ELIGIBILITY:
Inclusion Criteria:

* Age between 15-80 years (US only), and 18-80 (rest of world (ROW)), male or female.
* Adjuvant or neoadjuvant chemotherapy (including doxorubicin) allowed if no tumor recurrence for at least 12 months since the last measurement, beginning or end of last chemotherapy.
* Histologically or cytologically confirmed, locally advanced, unresectable, and/or metastatic soft tissue sarcoma of intermediate or high grade.
* Capable of providing informed consent and complying with trial procedures.
* ECOG performance status 0-2.
* Life expectancy > 12 weeks.
* Measurable tumor lesions according to RECIST 1.1 criteria.
* Women must not be able to become pregnant (e.g. post-menopausal for at least 1 year, surgically sterile, or practicing adequate birth control methods) for the duration of the study. (Adequate contraception includes: oral contraception, implanted contraception, intrauterine device implanted for at least 3 months, or barrier method in conjunction with spermicide.)
* Women of child bearing potential must have a negative serum or urine pregnancy test at the Screening Visit and be non-lactating.
* Geographic accessibility to the site that ensures the subject will be able to keep all study-related appointments.

Exclusion Criteria:

* Prior chemotherapy unless for adjuvant or neoadjuvant therapy with no tumor recurrence for at least 12 months.
* Prior exposure to > 3 cycles or 225 mg/m2 of doxorubicin or Doxil®.
* Palliative surgery and/or radiation treatment less than 4 weeks prior to Randomization.
* Exposure to any investigational agent within 30 days of Randomization.
* Current Stage 1 or 2 soft tissue sarcomas.
* Current evidence/diagnosis of alveolar soft part sarcoma, chondrosarcoma, rhabdomyosarcoma, osteosarcoma, gastrointestinal stromal tumor (GIST), dermatofibrosarcoma, Ewing's sarcoma, Kaposi's sarcoma, mixed mesodermal tumor, clear cell sarcomas and unresectable low grade liposarcomas.
* Central nervous system metastasis
* History of other malignancies except cured basal cell carcinoma, superficial bladder cancer or carcinoma in situ of the cervix unless documented free of cancer for > 5 years.
* Laboratory values: Screening serum creatinine > 1.5x upper limit of normal (ULN), alanine aminotransferase (ALT) > 3 × ULN or >5 × ULN if liver metastases are present, total bilirubin > 3 × ULN, absolute neutrophil count < 1,500/mm3, platelet concentration < 100,000/mm3, hematocrit level < 25% for females or < 27% for males, or coagulation tests (prothrombin time [PT], partial thromboplastin time [PTT], International Normalized Ratio [INR]) > 1.5 × ULN, albumin < 2.0 g/dL.
* Clinically evident congestive heart failure > class II of the New York Heart Association (NYHA) guidelines.
* Current, serious, clinically significant cardiac arrhythmias, defined as the existence of an absolute arrhythmia or ventricular arrhythmias classified as Lown III, IV or V.
* Baseline QTc > 470 msec and/or previous history of QT prolongation while taking other medications. Concomitant use of medications associated with a high incidence of QT prolongation is not allowed.
* History or signs of active coronary artery disease with or without angina pectoris.
* Serious myocardial dysfunction defined as scintigraphically (e.g. MUGA, myocardial scintigram) or ultrasound determined absolute left ventricular ejection fraction (LVEF) < 45% of predicted.
* History of HIV infection.
* Active, clinically significant serious infection requiring treatment with antibiotics, anti-virals or anti-fungals.
* Major surgery within 3 weeks prior to Randomization.
* Substance abuse or any condition that might interfere with the subject's participation in the study or in the evaluation of the study results.
* Any condition that is unstable and could jeopardize the subject's participation in the study.

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2012-01-11 (Actual); Primary Completion 2014-04-09 (Actual); Study Completion 2014-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sant Chawla, M.D., Principal Investigator — Sarcoma Oncology Center; Daniel Levitt, M.D., Ph.D., Study Director — CytRx
Locations (34):
- United States (5):
  - Sarcoma Oncology Center, Santa Monica, California
  - Stanford University, Stanford, California
  - University of Iowa, Iowa City, Iowa
  - Pennsylvania Hematology Oncology Associates, Philadelphia, Pennsylvania
  - CTRC Institute for Drug Development, University of Texas, San Antonio, Texas
- Australia (7):
  - Royal North Shore, St Leonards, New South Wales
  - Epworth HealthCare Clinical Trials and Research Centre, Richmond, Victoria
  - Border Medical Oncology, Wodonga, Victoria
  - Royal Hobart Hospital, Hobart
  - Royal Perth Hospital, Perth
  - Mount Medical Centre, Perth
  - The Crown Princess Mary Cancer Centre Westmead, Sydney
- State Health Centre Oncology Department, Budapest, Hungary
- India (10):
  - Hemato Oncology Clinic, Vedanta Institute of Medical Science, Thaltej, Ahmedaba
  - Hemato Oncology Clinic, Vedanta Institute of Medical Science, Ahmedabad, Gujarat
  - M.S. Ramaiah Medical College and Hospitals, Bangalore, Karnataka
  - Curie Manavata Cancer Centre, Nashik, Maharashtra
  - Delhi State Cancer Institute, Pune, Maharashtra
  - Jehangir Clinical Development Centre Pvt Ltd, Pune, Maharashtra
  - Delhi State Cancer Institute, Mandoli, National Capital Territory of Delhi
  - Noble Hospital Clinical Research Department 1st Floor, Hadapsar, Pune Maharashtra
  - Christian Medical College, Vellore, Tami Nadu
  - Tata Memorial Hospital, Department of Medical Oncology, Mumbai
- Romania (4):
  - Oncological Institute "Prof. Dr. I. Chiricuta", Cluj-Napoca, Cluj-Napoca, County Cluj
  - Clinical County Hospital Mures, Medical Oncology Department, Târgu Mureş, County Mures
  - Spitalul Judetean de Urgenta "Dr. Constantin Opris" Baia-Mare, Sectia Oncologie, Baia Mare, Judet Maramures
  - Medisprof SRL, Cluj-Napoca
- Russia (2):
  - State Healthcare Institution "Republican Clinical Oncological Center of the Ministry of Health of Republic of Tatarstan", Kazan', Tatarstan Republic
  - Blokhin Cancer Research Center, Moscow
- Ukraine (5):
  - Municipal institution "Chernivtsi Regional Clinical Oncologic Dispensary",, Chernivtsi
  - Municipal Institution "Dnipropetrovsk City Multi-Field Clinical Hospital #4" of Dnipropetrovsk Regional Councel, Dnipropetrovsk
  - State Institution "Institute of Medical Radiology named after S.P.Grygoryev of National Academy of Medical Sciences of Ukraine",, Kharkiv
  - Lviv State Oncological Regional Treatment - Diagnostics Center, Chemotherapy Department, Lviv
  - Vinnytsya Regional Clinical Oncologic Dispensary, Surgical Department, Vinnytsia

REFERENCES:
- [Derived] Chawla SP, Papai Z, Mukhametshina G, Sankhala K, Vasylyev L, Fedenko A, Khamly K, Ganjoo K, Nagarkar R, Wieland S, Levitt DJ. First-Line Aldoxorubicin vs Doxorubicin in Metastatic or Locally Advanced Unresectable Soft-Tissue Sarcoma: A Phase 2b Randomized Clinical Trial. JAMA Oncol. 2015 Dec;1(9):1272-80. doi: 10.1001/jamaoncol.2015.3101. PMID 26378637
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/26378637/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/25312684/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 126 subjects were randomized to the intent to treat population, whereas 123 were in the safety population.
  3 subjects were randomized, but not treated.
Groups:
- Doxorubicin: Doxorubicin: Doxorubicin administered at 75 mg/m^2 for up to 6 consecutive cycles.
- INNO-206: INNO-206: INNO-206 administered at 350 mg/m^2 (260 mg/m^2 doxorubicin equivalent) intravenously (IV) on Day 1 every 21 days for up to 6 consecutive cycles
Period: Overall Study
Arm/Group | Doxorubicin | INNO-206
Started | 40 | 83
Completed | 17 | 50
Not Completed | 23 | 33
Not completed — Adverse Event | 3 | 5
Not completed — Withdrawal by Subject | 2 | 4
Not completed — Protocol Violation | 2 | 4
Not completed — Physician Decision | 0 | 2
Not completed — Disease Progression | 13 | 14
Not completed — Death | 1 | 3
Not completed — Other | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Doxorubicin | INNO-206 | Total
Number analyzed (Participants) | 40 | 83 | 123
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.5 (12.42) | 52.3 (13.91) | 53 (13.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 45 | 67
  Male | 18 | 38 | 56
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 16 | 22
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 1 | 1 | 2
  White | 32 | 61 | 93
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 5 | 5
Subjects with Metastatic, Locally Advanced, or Unresectable Soft Tissue Sarcoma [Count of Participants; unit: Participants] | 40 | 83 | 123

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Progression-free survival is defined as the interval from the date of registration (ie, assignment of subject number) to the earliest date of documented evidence of recurrent or progressive disease, or the date of death due to any cause, whichever occurs first.
  Progressive Disease is defined as: 20% increase in the sum of the longest diameter of target lesions from the smallest sum of the longest diameter recorded since the treatment started; the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of 1 new lesion is also considered progression.
Time Frame: Approximately 24 months
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Doxorubicin | INNO-206
Number analyzed (Participants) | 40 | 83
Days | 83 [48 to 132] | 170 [92 to 246]

2. Secondary Outcome: Overall Survival
Description: Overall survival was measured from the date of registration (ie, assignment of subject number) to the date of death due to any cause, or the date of last contact.
Time Frame: Approximately 35 months
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Doxorubicin | INNO-206
Number analyzed (Participants) | 40 | 83
Days | 434 [261 to 627] | 480 [394 to NA] — The upper 95% Confidence Interval was not reached.

3. Secondary Outcome: Progression-free Survival at 4 and 6 Months
Time Frame: Month 4 and 6
Population: 126 subjects were randomized to the intent to treat population, whereas 123 were in the safety population.
  3 subjects were randomized, but not treated.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Doxorubicin | INNO-206
Number analyzed (Participants) | 38 | 80
percentage of participants
  Percentage of participants at 4 Months (%) | 40.8 [24.5 to 56.5] | 60 [47.9 to 70.1]
  Percentage of participants at 6 Months (%) | 22.9 [10.0 to 38.9] | 45.7 [33.7 to 57.0]

4. Secondary Outcome: Objective Overall Response Rate (ORR)
Description: Objective Overall Response will be evaluated using the Response Evaluation Criteria In Solid Tumors 1.1 (RECIST 1.1). Changes (i.e., improvements) in tumor measurements from baseline values will be assigned a status of CR or PR. Objective response measurements will comprise the sum of CR plus PR.
  Complete Response (CR): disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm).
  Partial Response (PR): 30% decrease in the sum of the longest diameter of target lesions, from the baseline sum longest diameter.
Time Frame: Approximately 24 months
Measure: Number (95% Confidence Interval); unit: Percentage of Subjects
Arm/Group | Doxorubicin | INNO-206
Number analyzed (Participants) | 38 | 80
Percentage of Subjects | 0 [0 to 9.3] | 25 [16 to 35.9]

5. Secondary Outcome: Number of Participants With Treatment-related Toxicities (Adverse Events)
Description: Treatment will continue every 21 days until tumor progression is observed, 6 cycles of treatment are completed or unacceptable toxicity occurs.
Time Frame: 30 days after last dose, up to 136 days (6 cycles of treatment plus 30 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Doxorubicin | INNO-206
Number analyzed (Participants) | 40 | 83
Participants | 29 | 75

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) that occurred after any administration of the study medication were to be followed until the event resolved, until the subject began alternative treatment, or until 30 days after the last dose of study medication. All SAEs that occurred during the course of the study or within 30 days of the last administration of study medication were to be reported. 30 days after last dose, up to 136 days (6 cycles of treatment plus 30 days).
Arm/Group | Doxorubicin | INNO-206
All-Cause Mortality (participants affected / at risk) | 26/40 | 40/83
Serious Adverse Events (participants affected / at risk) | 8/40 | 33/83
Other Adverse Events (participants affected / at risk) | 32/40 | 79/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Doxorubicin (N=40) | INNO-206 (N=83)
Febrile Neutropenia (Blood and lymphatic system disorders) | 5 | 11
Anaemia (Blood and lymphatic system disorders) | 3 | 6
Leukopenia (Blood and lymphatic system disorders) | 0 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 2
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 2
Vomiting (Gastrointestinal disorders) | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 3
Pneumonia (Infections and infestations) | 1 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Neutropenic sepsis (Infections and infestations) | 0 | 1
Oral herpes (Infections and infestations) | 0 | 1
Pertussis (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 1 | 0
Tooth infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Pyrexia (General disorders) | 0 | 3
Mucosal inflammation (General disorders) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 2
Hypovolaemic shock (Vascular disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Atrial tachycardia (Cardiac disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Pelvic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Doxorubicin (N=40) | INNO-206 (N=83)
Nausea (Gastrointestinal disorders) | 11 | 38
Stomatitis (Gastrointestinal disorders) | 5 | 28
Vomiting (Gastrointestinal disorders) | 7 | 19
Constipation (Gastrointestinal disorders) | 2 | 12
Diarrhoea (Gastrointestinal disorders) | 7 | 7
Abdominal Pain (Gastrointestinal disorders) | 2 | 8
Anaemia (Blood and lymphatic system disorders) | 13 | 36
Neutropenia (Blood and lymphatic system disorders) | 7 | 33
Febrile neutropenia (Blood and lymphatic system disorders) | 7 | 13
Leukopenia (Blood and lymphatic system disorders) | 4 | 15
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 12
Fatigue (General disorders) | 6 | 24
Asthenia (General disorders) | 5 | 15
Pyrexia (General disorders) | 3 | 14
Mucosal inflammation (General disorders) | 2 | 10
Oedema peripheral (General disorders) | 3 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 12 | 25
Decreased appetite (Metabolism and nutrition disorders) | 2 | 20
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 8
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 8
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 9
Aspartate aminotransferase increased (Investigations) | 3 | 6
Weight decreased (Investigations) | 2 | 7
Blood alkaline phosphatase increased (Investigations) | 1 | 7
Alanine aminotransferase increased (Investigations) | 2 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 5
Ejection fraction decreased (Investigations) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-04-15): https://cdn.clinicaltrials.gov/large-docs/88/NCT01514188/Prot_SAP_000.pdf